CLINICAL TRIAL: NCT05760573
Title: Ready and Healthy for Kindergarten: A Primary Care Innovation to Promote a 360-degree View of Child Health
Brief Title: The Ready and Healthy for Kindergarten Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Associate Professor of Pediatrics & Family Medicine and Community Health, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2021001575-2; R18HS028574 (AHRQ)
Record Dates: First submitted 2023-02-04; First posted 2023-03-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Parenting; Language Development; Literacy; Health Behavior
Keywords: early literacy; language development; famliy literacy; bilingualism; community engagement
MeSH Terms: conditions — Literacy; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care plus school supplies and resources (No Intervention): This group will not be enrolled in the Family Wellness Program. They will receive usual care from their regular clinician plus a backpack with schools supplies and a list of resources.
- Famliy Wellness Program (Experimental): This group will be enrolled in the Family Wellness Program which consists of 8 weekly parent-child workshops prior to the children entering kindergarten as well as 4 booster sessions during the child's kindergarten year. As part of the program families will receive school supplies, books and resources.
  Interventions: Behavioral: Family Wellness Program (FWP)

INTERVENTIONS:
Behavioral: Family Wellness Program (FWP) — The FWP will consist of the following general format: (1) 8 weekly 60-minute summer workshops; (2) 4 booster workshops throughout the year; and (3) 2-3 outreach text messages per week for 10 months.
  Arms: Famliy Wellness Program

SUMMARY:
The goal of this clinical trial is to test whether a family wellness program enhances child and parenting outcomes among Latino dual language learners entering Kindergarten and their families. The main questions are: (1) To what extent does the family wellness program enhance home health and learning routines, and (2) To what extent does the family wellness program enhance child literacy, language, and social-emotional outcomes.

All participants will be asked to complete surveys and assessments.

Researchers will compare two groups: (1) Family wellness program that includes (a) 8-weekly summer sessions, (b) text messages, (c) booster sessions, and (2) usual care plus school supplies and list of resources to see if the family wellness program enhances child and parenting outcomes.

DETAILED DESCRIPTION:
Education is a critical social determinant of health (SDOH). Latino dual language learners face large gaps in school readiness, which perpetuate inequities in academic achievement and subsequent health. Investigators developed an online family wellness program that uses anticipatory guidance on health topics intrinsically important to school readiness (e.g., nutrition, physical activity) to introduce basic language and literacy skills to Latino dual language learners, a fast- growing and particularly high-risk group, and their families. The online family wellness program was developed through a cross-sector partnership between educators and pediatric professionals and consists of parent-child workshops and reminder text messages. The program occurs during the transition into Kindergarten, a critical developmental stage, and uses promising approaches such as group structure, strategic use of technology, and partnerships. The program tightly integrates Bright Futures anticipatory guidance with the Kindergarten curriculum. During pilot testing, the investigators found that the family wellness program was feasible, well attended, and highly acceptable. The investigators now propose testing the effect of the family wellness program on child and parenting outcomes using a rigorous mixed methods and community-engaged approach. The investigators will conduct a randomized controlled trial testing the effects of the family wellness program on child language, literacy, and social-emotional outcomes as well home health and learning routines. The investigators will also conduct a mixed methods process evaluation, which will provide insight into reach and implementation as well as user experience.

ELIGIBILITY:
Inclusion Criteria:

* primary caregiver of a child entering Kindergarten (4-6 years old),
* primary caregiver identifies as Hispanic/Latino/Latinx,
* family speaks Spanish at home,
* cell phone ownership,
* willing to receive text messages,
* ability to pick up program materials locally, and
* willing to accept randomization

Exclusion Criteria:

-Individuals unable to provide informed consent

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Home Literacy Environment Questionnaire | 2 months
  The home literacy environment will be assessed with the StimQ, a caregiver-reported measure of cognitive stimulation for children that includes a domain on the home literacy environment (READ scale). The READ scale includes 3 subdimensions (Book Reading Quantity, Diversity of Content, Book Reading Quality). Scores on the READ scale range from 0 to 18. Higher scores indicate more cognitive stimulation
Home Literacy Environment Questionnaire | 10 months
  The home literacy environment will be assessed with the StimQ, a caregiver-reported measure of cognitive stimulation for children that includes a domain on the home literacy environment (READ scale). The READ scale includes 3 subdimensions (Book Reading Quantity, Diversity of Content, Book Reading Quality). Scores on the READ scale range from 0 to 18. Higher scores indicate more cognitive stimulation
Parent Responsiveness Questionnaire | 2 months
  Parent responsiveness will be assessed with the StimQ, a caregiver-reported measure of cognitive stimulation for children that includes a domain on responsiveness (Parental Verbal Responsiveness scale). The Parental Verbal Responsiveness scale includes a subdimension on responsiveness during routines (Everyday Routines). Scores range from 0 to 8. Higher scores indicate more cognitive stimulation.
Parent Responsiveness Questionnaire | 10 months
  Parent responsiveness will be assessed with the StimQ, a caregiver-reported measure of cognitive stimulation for children that includes a domain on responsiveness (Parental Verbal Responsiveness scale). The Parental Verbal Responsiveness scale includes a subdimension on responsiveness during routines (Everyday Routines). Scores range from 0 to 8. Higher scores indicate more cognitive stimulation.
Family Health Routines Questionnaire | 2 months
  This is a self-report measure for family nutrition and physical activity routines, which has been validated in English and Spanish. Higher scores are consistent with healthier routines.
Family Health Routines Questionnaire | 10 months
  This is a self-report measure for family nutrition and physical activity routines, which has been validated in English and Spanish. Higher scores are consistent with healthier routines.
Caregiver Attitudes About Reading Questionnaire | 2 months
  The Parent Reading Belief Inventory is a caregiver reported measure of attitudes and knowledge about reading with children that includes subdimensions of teaching efficacy (scores range from 0 to 27), positive affect (scores range from 0 to 33), and knowledge (scores range from 0 to 15) available in English and Spanish. Higher scores indicate more favorable attitudes and greater knowledge.
Caregiver Attitudes About Reading Questionnaire | 10 months
  The Parent Reading Belief Inventory is a caregiver reported measure of attitudes and knowledge about reading with children that includes subdimensions of teaching efficacy (scores range from 0 to 27), positive affect (scores range from 0 to 33), and knowledge (scores range from 0 to 15) available in English and Spanish. Higher scores indicate more favorable attitudes and greater knowledge.
Child Vocabulary Assessment | 2 months
  Child vocabulary will be assessed using an investigator developed measure. Higher scores indicate higher skills
Child Vocabulary Assessment | 10 months
  Child vocabulary will be assessed using an investigator developed measure. Higher scores indicate higher skills
Child Language Skills Assessment | 10 months
  Child receptive language and listening skills will be assessed with the Receptive One Word Picture Vocabulary Test - Fourth Edition (ROWPVT-4) Spanish-Bilingual. Higher scores indicate higher skills.
Child Literacy Skills Assessment | 2 months
  Literacy skills including concepts about books, story retelling, narrative thematic knowledge, letter and sound identification will be assessed using an investigator developed measure. Higher scores indicate higher skills
Child Literacy Skills Assessment | 10 months
  Literacy skills including concepts about books, story retelling, narrative thematic knowledge, letter and sound identification will be assessed using an investigator developed measure. Higher scores indicate higher skills
Child Social-emotional Development Questionnaire | 2 months
  Social emotional development will be measured using the Strengths and Difficulties Questionnaire (SDQ), which is a brief validated behavioral screening questionnaire for 4-17 year olds. The SDQ has been widely used in research studies. The SDQ has a total of 5 scales including the hyperactivity (scores range from 0-10) and prosocial (scores range from 0-10) scales used here. Higher scores on the hyperactivity scale indicate greater hyperactivity; higher scores on the Prosocial scale indicate greater prosocial behaviors.
Child Social-emotional Development Questionnaire | 10 months
  Social emotional development will be measured using the Strengths and Difficulties Questionnaire (SDQ), which is a brief validated behavioral screening questionnaire for 4-17 year olds. The SDQ has been widely used in research studies. The SDQ has a total of 5 scales including the hyperactivity (scores range from 0-10) and prosocial (scores range from 0-10) scales used here. Higher scores on the hyperactivity scale indicate greater hyperactivity; higher scores on the Prosocial scale indicate greater prosocial behaviors.

SECONDARY OUTCOMES:
Child Media Use Questionnaire | 2 months
  The ScreenQ is a caregiver report measure of media use in children. Scores range from 0 to 26 with higher score indicating more media use.
Child Media Use Questionnaire | 10 months.
  The ScreenQ is a caregiver report measure of media use in children. Scores range from 0 to 26 with higher score indicating more media use.
Child Sleep Routines Questionnaire | 2 months
  Investigator developed question on sleep habits.
Child Sleep Routines Questionnaire | 10 months
  Investigator developed question on sleep habits.
Child Self-regulation Questionnaire | 2 months
  Using observational method by using a popular children's song to measure child's self regulation.
Child Self-regulation Questionnaire | 10 months
  Using observational method by using a popular children's song to measure child's self regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel E Jimenez, MD, MS, Principal Investigator — Rutgers University
Locations (1):
- Child Health Institute, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified quantitative data and associated documentation may be made available to users conducting non-profit research under a written data-sharing agreement
Supporting Information: Study Protocol
Time Frame: Data will become available after the study is completed and primary study findings are published in peer-reviewed journals for up to 10 years after study completion.
Access Criteria: Researchers from accredited institutions may submit written requests to access de-identified quantitative data for non-profit research. Permission and access will be granted on an ad hoc basis and under a written data-sharing agreement. The dataset will be stripped of all identifiers prior to sharing and will be shared via a secure application.